CLINICAL TRIAL: NCT03424252
Title: A Phase 1, Open-label, Crossover, Randomised Study to Evaluate the Pharmacokinetic Profile of FDL169 Sublingual Formulations in the Fed State in Healthy Subjects
Brief Title: An Phase 1 Study to Evaluate the Pharmacokinetic (PK) Profile of FDL169 New Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Flatley Discovery Lab LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FDL169-2017-05
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FDL169 Dose Level 1,sublingual to oral (Experimental): Dose level 1 sublingual first and oral second.
  Interventions: Drug: FDL169
- FDL169 Dose Level 1 dosing,oral to sublingual (Experimental): Dose level 1 oral first and sublingual second.
  Interventions: Drug: FDL169
- FDL169 Dose Level 2 sublingual to oral,Optional (Experimental): Dose level 2 sublingual first and oral second.
  Interventions: Drug: FDL169
- FDL169 Dose Level 2 oral to sublingual,Optional (Experimental): Dose level 2 oral first and sublingual second.
  Interventions: Drug: FDL169

INTERVENTIONS:
Drug: FDL169 — Cystic Fibrosis Transmembrane Regulator (CFTR) corrector

SUMMARY:
Two parts, two periods, crossover study with part 2 is optional. In both parts, subjects will be randomized to sequentially receive both sublingual and oral formulations of FDL169.

DETAILED DESCRIPTION:
This is a single center, open label study on healthy volunteers. The study will consist of up to 2 parts; the decision to proceed to the optional second part will be made following review of Part 1 data. Part 1 and optional Part 2 have randomized, 2 period crossover designs. Subjects will randomized to 1 of 2 treatment sequences in order to receive 2 single doses of FDL169 on separate occasions, one as a sublingual administration and one as an oral administration. There will be a minimum washout period of 10 days between FDL169 administrations. The duration of each part is approximately 7 weeks from screening to follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females
2. Body mass index of 18.0 to 32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
3. Must agree to follow the study's contraception requirement Subject has normal healthy oral mucosa with no clinically significant findings

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the previous 3 months
2. Subjects who have previously received FDL169
3. History of any drug or alcohol abuse in the past 2 years
4. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
5. Current smokers and those who have smoked within the last 12 months
6. Females of childbearing potential who are pregnant or lactating (all female subjects must have a negative urine pregnancy test at screening and each admission). A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy) or is postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle-stimulating hormone [FSH] concentration >40 mIU/mL)
7. Alkaline phosphatase, aspartate aminotransferase and/or alanine aminotransferase level >1.5 x upper limit of normal at screening
8. Abnormal renal function at screening, defined as estimated glomerular filtration rate <60 mL/min using the Modification of Diet in Renal Disease (MDRD) equation
9. Clinically significant abnormal biochemistry, haematology, coagulation or urinalysis as judged by the investigator (laboratory parameters are listed in)
10. Positive drugs of abuse test result
11. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
12. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
13. Subjects with a history of abdominal surgery eg cholecystectomy (appendectomy is allowed unless procedure was within 12 months)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters, Cmax | 7 weeks
  The pharmacokinetic parameters of FDL169; maximal plasma concentration (Cmax)
Pharmacokinetic parameters, Tmax | 7 weeks
  The pharmacokinetic parameters of FDL169; maximal concentration (Tmax)
Pharmacokinetic parameters, AUC | 7 weeks
  The pharmacokinetic parameters of FDL169; area under the plasma concentration curve (AUC)
Pharmacokinetic parameters, CL/F | 7 weeks
  The pharmacokinetic parameters of FDL169; clearance (CL/F)
Pharmacokinetic parameters, V/F | 7 weeks
  The pharmacokinetic parameters of FDL169; apparent volume of distribution (V/F)
Ratio of pharmacokinetic parameters, AUC, between sublingual and oral formulation | 7 weeks
  The pharmacokinetic parameters of FDL169; area under the plasma concentration curve (AUC) of FDL169 and its M1 metabolite following sublingual dosing compared to oral dosing

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 7 weeks
  Safety and tolerability of FDL169 as determined by the incidence of adverse events (Aes) and serious adverse events (SAE)s.

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom